CLINICAL TRIAL: NCT03291119
Title: To Evaluate the Predictors of Risk Factors for Extubation Failure After Cervico-Vertebral Junction Surgery-A Prospective Observational Study.
Brief Title: Risk Predictors of Extubation Failure for Cervico-medullary Junction Surgery
Acronym: CVJ-RISK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Kiran Jangra, Principle Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: CVJ-RISK; NK/3172/Res/97 (Other: PGIMER)
Record Dates: First submitted 2017-03-06; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cervical Lesion
Keywords: Cervico-medullary, Extubation Failure, Risk Predictors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CVJ anomalies affecting skeleton might lead to the pressure on the neuraxis, and disturbance of the cerebrospinal fluid circulation and blood supply. The patients undergoing surgeries on CVJ might develop airway complications in immediate postoperative period warranting urgent reintubation or emergency tracheostomy. Reintubation is usually difficult in immediate postoperative period due the fixation of cervical spine and gross upper airway oedema due to prolonged surgery in prone position. This will be the first prospective observational study to find out the risk factors related to patient, anaesthesia, radiological findings and surgical procedure to predict extubation failure in patients undergoing CVJ surgeries.

DETAILED DESCRIPTION:
Research Query We conducted a pilot study and found that the incidence of reintubation is 20%. Reintubation poses a clinical, psychological and financial burden on the patients. Consequently, our study aims to identify the various risk factors to predict the need for reintubation and postoperative mechanical ventilation so that success of extubation can be anticipated.

Introduction:

The craniovertebral junction (CVJ) includes the basiocciput, atlas, axis and various supporting ligaments. The contents enclosed in CVJ include Medulla, cervical spinal cord (cervico-medullary junction), spinal arteries, and lower cranial and cervical nerves1. CVJ anomalies affecting skeleton might lead to the pressure on the neuraxis and disturbance of the cerebrospinal fluid circulation and blood supply. The clinical manifestations of CVJ abnormalities include weakness of both upper and lower limbs, respiratory dysfunction due to compression of the respiratory centres in brainstem and weakness of respiratory muscles including diaphragm2. The patients undergoing surgeries on CVJ might develop airway complications in immediate postoperative period warranting urgent reintubation or emergency tracheostomy3. Reintubation is usually difficult in immediate postoperative period in the view of fixation of cervical spine and gross upper airway oedema due to prolonged surgery in prone position4,5. To avoid such airway emergencies few centres favour to delay the extubation. The patients with weak respiratory muscles and poor respiratory reserve tend to develop major pulmonary complications and become ventilator dependant so, we always plan an early weaning and extubation6-9.

Epstein et al10 reported that the potential risk factors associated with postoperative emergency airway management following cervical spine surgery included; obesity (>220 ponds), surgery duration greater than 10 hours, anterior corpectomy with fusion of second cervical vertebra, greater than 4 units of transfused blood, asthma, advanced age (>65 years), a cerebrospinal fluid fistula, extent surgery, and severe preoperative neurologic deficit. These risk factors are generalised for all cervical surgeries. CVJ is an important area where most of the vital centres present in medulla are at risk of injuries that leads to central respiratory depression and even sudden death. These patients can have airway and respiratory compromise even in the absence of the risk factors described by Epstein et al10. Hence, we plan to conduct this study to identify the risk factors leading to extubation failure in patients undergoing surgeries for CVJ anomalies, so that, early or delayed extubation can be planned before the end of surgery.

NOVELTY:

This will be the first prospective observational study to find out the risk factors related to patient, anaesthesia, radiological findings and surgical procedure to predict extubation failure in patients undergoing CVJ surgeries. This will help in planning and predicting postsurgical extubation and psychological preparation of the patients who will need postoperative mechanical ventilation.

Relevance of Research Proposal to Public Health and in Given Area:

Both extubation failure and ventilatory dependence are the common problems and contribute significantly to the mortality and morbidities in the patients with CVJ surgeries. Till date we do not have specific parameters to predict the risk of extubation failure resulting in life threatening emergency situation during extubation of these patients. With this research, we might find certain risk factor that can clearly predict extubation failure and patients with those risk factors can be electively ventilated or tracheostomised.

Review of Literature The CVJ anomalies might lead to the compression on the vital neural structures and disturbance in cerebrospinal fluid circulation and blood supply1. These patients manifest with the weakness of both upper and lower limbs, respiratory muscles weakness or central suppression of ventilation2. These surgeries on CVJ might lead to airway complications in immediate postoperative period warranting urgent reintubation or emergency tracheostomy3. Reintubation is usually difficult in immediate postoperative period in the view of fixation of cervical spine and gross upper airway oedema due to prolonged surgery in prone position4,5. To avoid such airway emergencies few centres favour to delay the extubation. The patients with weak respiratory muscles and poor respiratory reserve tend to develop major pulmonary complications and become ventilator dependant so, we always plan an early weaning and extubation6-9.

National data on the CVJ surgeries Marda et al10 hypothesize that the respiratory system is compromised and sub-clinical manifestations may get aggravated postoperatively due to the anesthetic or surgical reasons. They evaluated the incidence of postoperative pulmonary complications (PPCs) and associated risk factors in patients undergoing combined procedure for transoral odontoidectomy (TOO) and posterior fixation (PF). The authors concluded that the patients with CVJ anomaly are at increased risk of developing PPCs and there is a strong association between intraoperative blood transfusion and PPCs. They also found that the patients PPCs had a longer ICU and hospital stay.

In another study, Marda et al11 compared the early and late extubation following transoral odontoidectomy and posterior fixation. They concluded that ventilation and oxygenation was comparable between the groups but the duration of ICU and hospital stay was prolonged in the delayed extubation group.

Reddy et al12 evaluated the pulmonary function after surgery for congenital atlantoaxial dislocation and compared with compressive myelopathy and cerebellar surgeries. The authors concluded that a significant deterioration of pulmonary function that persists till one week after surgery for congenital AAD and this deterioration was significantly higher than that seen after surgeries for compressive myelopathies and cerebellar lesion.

International Data on the CVJ surgeries Epstein et al13 reported that the potential risk factors associated with postoperative emergency airway management following cervical spine surgery included; obesity (>220 ponds), surgery duration greater than 10 hours, anterior corpectomy with fusion of second cervical vertebra, greater than 4 units of transfused blood, asthma, advanced age (>65 years), a cerebrospinal fluid fistula, extent surgery, and severe preoperative neurologic deficit.

These risk factors are generalised for all cervical surgeries. CVJ is an important area where most of the vital centres present in medulla are at risk of injuries that leads to central respiratory depression and even sudden death. These patients can have airway and respiratory compromise even in the absence of the risk factors described by Epstein et al13. Hence, we plan to conduct this study to identify the risk factors leading to extubation failure in patients undergoing surgeries for CVJ anomalies, so that, early or delayed extubation can be planned before the end of surgery.

Objectives:

Primary Objective:

To evaluate the predictors of extubation failure in patients undergoing surgeries for CVJ anomalies.

Secondary Objective:

To determine the association of various predictors with

1. Duration of postoperative mechanical ventilation
2. Duration of ICU stay
3. Duration of Hospital Stay
4. mortality

Preliminary work: We have done 10 pilot cases that shows reintubation rate of 20%. Rest of the data is yet to be analysed.

Research Design/Methodology:

This Prospective Observational study will be commenced after taking approval from Institutional Ethics committee and patients consent. A total of hundred patients will be enrolled.

Inclusion Criterion:

Patients with CVJ Anomalies posted for surgery

Exclusion Criterion:

1. Patients requiring preoperative intubation and ventilator support
2. Patients with

   1. Severe cardiac and pulmonary disease
   2. Morbid obesity
   3. Obstructive sleep apnoea
   4. Clinically significant scoliosis
   5. Severe neurological disability The "Extubation Failure" will be defined as inability to extubate within 24 hours or reintubation within 24 hours. Early extubation failure will be reintubation within 6 hours postoperatively and late extubation failure will be after 6 hours postoperatively.

The criteria for reintubation will include desaturation (PaO2 <60), hypoventilation (PaCO2 >50), tachypnea (RR >35/min), impending respiratory failure, stridor and retention of secretion.

Besides routine preoperative investigations respiratory reserve will be evaluated by room air Arterial Blood Gas analysis, Pulmonary function tests, Chest expansion and Breath holding time. These parameters will be repeated after 3 months on follow up. Neurological status will be assessed by using Benzel's modification of Japanese Orthopedic Association scoring system (mJOA score) 11 (Annexure-I).

Standard fasting protocol will be followed. Anaesthesia and intubation techniques and monitoring will be as per attending anaesthesiologist's discretion but records of these techniques will be kept.

The following intraoperative clinical parameters will be recorded:

* Hemodynamic instability
* Total blood loss
* Amount and type of intravenous fluids
* Blood and blood products transfusion
* Total blood loss
* Intraoperative complications such as vascular injuries/Dural tear Radiological abnormalities and dislocation axis will be noted. At the end of surgery patient will be reversed and assessed for possibility of extubation. Postoperative status will be evaluated. Patient will be followed up till discharge for any cardio-pulmonary events and three months later for assessment of pulmonary reserve.

ELIGIBILITY:
Lists of Inclusion Criterion

1.Patients with CVJ Anomalies posted for surgery

Lists of Exclusion Criterion:

1. Patients requiring preoperative intubation and ventilator support
2. Patients with Severe cardiac and pulmonary disease, Morbid obesity, Obstructive sleep apnoea, Clinically significant scoliosis, Severe neurological disability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CVJ Anomalies posted for surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-31 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Extubation failure will be evaluated in patients undergoing surgeries for CVJ surgery. | 1 year
  Extubation failure is defined as failure to extubate or reintubation with in 24 Hrs postoperatively.

SECONDARY OUTCOMES:
The association of various predictors with Outcome will be determined | 1 year
  Outcome is defined as Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Jangra, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No